CLINICAL TRIAL: NCT01957046
Title: A Single-arm, Open-label, Multicentre, Non-randomised, Study to Assess the Effect and Tolerability of Standardised Laxative Therapy for the Reversal of Opioid-induced Constipation in Subjects Suffering From Malignant or Non-malignant Pain That Requires Around-the-clock Opioid Therapy
Brief Title: A Single-arm, Study to Assess the Effect and Tolerability of Standardised Laxative Therapy (SLT) for the Reversal of Opioid-induced Constipation (OIC).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLT4501
Record Dates: First submitted 2013-07-10; First posted 2013-10-08 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Opioid Induced Constipation
Keywords: Opioid induced constipation; Laxatives
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — Laxatives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral Laxative (Other)
  Interventions: Drug: Laxative

INTERVENTIONS:
Drug: Laxative

SUMMARY:
The main purpose of this study is to assess how effective and tolerable the country specific clinical practice guidelines of SLTs are for UK, France and Sweden are.

The main rationale behind this study is that well controlled comparisons of the various laxatives for the treatment of OIC are lacking. There is lack of evidence suggesting which laxative or combination of laxatives is optimal for managing OIC.

DETAILED DESCRIPTION:
The study comprises of nine study visits and the total duration of the study is up to 42-52 days Potential subjects, aged 18 years and over, with OIC will be screened for entry into the study at Visit 1 Eligible subjects will attend a 7-day Screening Period (Visit 1). This will be followed by a 28-day Treatment Period (visits 2 to 8:), made up of four clinic visits scheduled 7 days apart (visits 5(day 7), 6(day 14), 7(day 21), 8(day 28): days 7 to 28) and two telephone visits (visits 3 and 4) which will take place during the first week of the Treatment Period. There will be a 7-day Follow-up Period with a follow-up phone call to conclude the study (Visit 9).

Study assessment/ evaluation include vital sign measurements, ECG, safety labs, pregnancy test and physical examination assessments, AEs, Investigator and subject questionnaires and subjects daily diaries.

Subjects will continue to take their prescribed pre-study opioid medication throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 18 years
* Females less than one year post-menopausal must have a negative pregnancy test prior to the first dose of study medication, be non-lactating, and willing to use adequate and highly effective methods of contraception throughout the study. (A highly effective method of birth control is defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly e.g. sterilisation, implants, injectables, combined oral contraceptives, some intrauterine devices ((IUDs), hormonal), sexual abstinence or vasectomised partner).
* Documented history of malignant or non-malignant pain that requires around-the-clock opioid therapy (WHO step II/III opioid analgesics).
* Subjects treated with WHO step II/III opioid analgesics for at least 2 weeks prior to Screening Visit (Visit 1), who will continue with the opioid(s) over the proposed study period.
* Subjects meeting the following criteria for OIC:

  * Subject and Investigator confirm that the Subject's constipation is induced, or worsened by the Subject's opioid medication (present at Screening)
  * Subjects with mean BFI score > 30 at Visit 1
  * Subjects with < 3 complete bowel movements (CBMs) in the week preceding the Visit 1, based on Subject's retrospective memory in response to Investigator's question.
* Subjects taking at least one laxative on regular basis (i.e. ≥2 intakes per week during the ≥2 weeks prior to screening) for the treatment of OIC.
* Subjects must be willing to take SLT.
* Subjects taking daily natural dietary fibre supplementation are eligible if they can maintain their diet throughout the study, and in the Investigator's opinion are willing and able to maintain adequate hydration.
* Subjects must be willing and able (e.g. mental and physical condition) to participate in all aspects of the study, including use of medication, completion of subjective evaluations, attending scheduled clinic visits, completing telephone contacts, and compliance with protocol requirements as evidenced by providing written, informed consent.
* In the Investigator's opinion the Subject's concomitant medication dose will remain stable throughout the study Period (here concomitant medications mean all medications besides opioids (standard and rescue opioid treatment)).

Exclusion Criteria:

Medical Conditions:

* In the Investigator's opinion any contraindication and precautionary condition for laxative medication(s) used in the study as per the SmPC.
* Subjects having any potential non-opioid cause of constipation that might be a major contributor.
* Surgery within 2 months prior to the start of the Screening Visit (Visit 1), or planned surgery during the Screening and Treatment periods that may affect GI motility.
* Subjects with colostomy or ileostomy.
* Hospitalisation expected/planned within the study Period (e.g. planned hospitalisation for the treatment of a pre-existing condition before informed consent) which can affect the outcome measure analysis.

Treatments/Medications:

• Subjects presently taking, or who have taken opioid antagonist(e.g. naloxone, naltrexone and methylnaltrexone) or opioid antagonists containing products (e.g. oxycodone/naloxone, buprenorphine/naloxone, pentazocine/naloxone, tilidine/naloxone) < 30 days prior to the start of the Screening Period.

* Subjects already taking maximum daily dose of country specific SLT (both First and Second Line SLT) on a regular basis (i.e. ≥4 days per week) for the treatment of OIC.
* Subjects receiving opioid substitution therapy for opioid addiction (e.g. methadone or buprenorphine).

Additional Screening Exclusion Criteria for Subjects Suffering from Non-malignant Pain:

- Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry

Additional Screening Exclusion Criteria for Subjects Suffering from Malignant Pain:

* Subjects who have received a new chemical entity or an experimental drug within 30 days of study entry (defined as Visit 1). Concurrent participation in another clinical trial is not permitted except the epidemiological study performed to assess the long-term survival data.
* Subjects with an expected life expectancy of < 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in soft complete bowel movements | Change from baseline
  Recorded in patient diary as and when occurs

SECONDARY OUTCOMES:
Change from baseline (Visit 2 to 8 (Day 1 to 28)) in SCBM - Non Straining | change from baseline
Additional laxative use (including enema) in addition to SLT (First Line and Second Line) | between visits and overall
Additional procedures (e.g. manual bowel evacuation or surgical procedure) required in addition to SLT | between visits and overall
Bowel Function Index (change from baseline to each visit (Day 7, 14, 21 and 28)) | change from baseline
Compliance with SLT/opioid therapy (premature discontinuation, SLT/opioid dose reduction or completely stopped SLT/opioid therapy). | from baseline to end of treatment
SLT/opioid-related AE and dropouts. | to end of treatment
The modified Subjective Opiate Withdrawal Scale at Day 7 and Day 28 | Day 7 and Day 28
The Clinical Opiate Withdrawal Scale at Day 7 and Day 28 | Day 7 and Day 28
Pain Intensity Scale - "Average Pain over last 24 Hours" at each visit (Day 7, 14, 21 and 28) | Day 7, 14, 21 and 28
The 36-item Short Form Health Survey (SF-36 v2) at Day 7 and Day 28 | Day 7 and 28
Clinical Global Impression (CGI) item 1 (severity) Day 28 | Day 28
Clinical Global Impression (CGI) item 2-4 (condition, therapeutic effect, side effects) Day 7 amd 28 | Day 7 and 28
The patient global impression of improvement (PGI-I) Day 28 | Day 28
Healthcare resources used for OIC treatment during the study (between first dose and last dose during the four week treatment period). | overall

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Support, Örebro, Sweden

REFERENCES:
- See also: Study Results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=SLT4501